CLINICAL TRIAL: NCT00436163
Title: Baltic Post-marketing Program of PEGASYS (Peg Interferon Alpha-2a 40KD) in Patients With HBeAg-positive and HBeAg-negative Chronic Hepatitis B
Brief Title: A Study of Peginterferon Alfa-2a (40KD) (PEGASYS®) in Participants With Hepatitis B Envelope Antigen (HBeAg) - Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20601
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon Alfa-2a (Experimental): Participants received peginterferon alfa-2a (Pegasys) 180 mcg subcutaneously once per week for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 mcg subcutaneously once per week for 48 weeks.
  Other Names: Pegasys®

SUMMARY:
This single-arm study will evaluate the efficacy and safety of peginterferon alfa-2a in treatment-naive Baltic participants with Hepatitis B envelope antigen (HBeAg)-positive chronic Hepatitis B virus (HBV). All participants will receive peginterferon alfa-2a 180 micrograms (mcg) subcutaneously once weekly. Following 48 weeks of treatment, there will be a 24 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is less than 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, 18-70 years of age;
* HBeAg positive, Hepatitis B surface antigen (HBsAg) positive for greater than or equal to 6 months;
* anti-HBs negative;
* Hepatitis B virus deoxyribonucleic acid (HBV DNA) greater than 5,00,000 copies/milliliters.

Exclusion Criteria:

* Previous antiviral or interferon-based therapy for chronic hepatitis B;
* Evidence of decompensated liver disease;
* Chronic liver disease other than viral hepatitis;
* Co-infection with active hepatitis A, C or D virus;
* Co-infection with human immunodeficiency virus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Estonia (2):
  - Tallinn
  - Tartu
- Riga, Latvia
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2a: Participants received peginterferon alfa-2a (Pegasys®) 180 micrograms (mcg) subcutaneously once per week for 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a
Started | 39
Completed | 36
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of peginterferon alfa-2a.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.28 (13.141)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Hepatitis B Envelope Antigen (HBeAg) Positive Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) Less Than (<) 1,00,000 Copies Per Milliliter (Copies/mL)
Description: HBeAg is a soluble antigen of hepatitis B virus present in the blood during acute infection, and disappear afterward but sometimes persisting in chronic disease. HBeAg positive participants were defined as those who had HBV DNA greater than (>) 1,00,000 copies/mL at baseline. This outcome measured the number of participants with HBV-DNA levels < 1,00,000 copies/mL at Week 72, who were defined as HBeAg positive at baseline.
Time Frame: Week 72
Population: All enrolled participants who received at least 1 dose of peginterferon alfa-2a. Here, Number of participants analyzed = participants who were HBeAg positive at baseline.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 22
participants | 6

2. Primary Outcome: Number of HBeAg Negative Participants With HBV-DNA < 10,000 Copies/mL
Description: HBeAg is a soluble antigen of hepatitis B virus present in the blood during acute infection, and disappear afterward but sometimes persisting in chronic disease. HBeAg negative participants were defined as those who had HBV DNA >10,000 copies/mL at baseline. This outcome measured the number of participants with HBV DNA <10,000 copies/mL at Week 72, who were defined as HBeAg negative at baseline.
Time Frame: Week 72
Population: All enrolled participants who received at least 1 dose of peginterferon alfa-2a. Here, Number of participants analyzed = participants who were HBeAg negative at baseline.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 17
participants | 6

3. Secondary Outcome: Number of Participants With HBV-DNA < 400 Copies/mL
Time Frame: Week 72
Population: All enrolled participants who received at least 1 dose of peginterferon alfa-2a. Here, Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 37
participants | 4

4. Secondary Outcome: Percentage of Hepatitis B Surface Antigen (HBsAg) Negative Participants
Description: HBsAg seroconversion was defined as the absence of HBsAg (HBsAg negative) and the presence of anti-HBs (anti-HBs positive) for HBsAg participants. Percentage of HBsAg negative participants were reported.
Time Frame: Week 48 and Week 72
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Peginterferon Alfa-2a: Participants received peginterferon alfa-2a (Pegasys)180 mcg subcutaneously once per week for 48 weeks.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 36
percentage of participants
  Week 48 | 3
  Week 72 | 3

5. Secondary Outcome: Percentage of Anti-HBs Positive Participants
Description: HBsAg seroconversion was defined as the absence of HBsAg (HBsAg negative) and the presence of anti-HBs (anti-HBs positive) for HbsAg participants. Percentage of Anti-HBs positive participants were reported.
Time Frame: Week 48 and Week 72
Population: All enrolled participants who received at least 1 dose of peginterferon alfa-2a. Here, Number of participants analyzed = participants evaluable for this outcome and n= participants with available data at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 36
percentage of participants
  Week 48 (n= 36) | 8
  Week 72 (n= 35) | 3

6. Secondary Outcome: Mean Alanine Aminotransferase (ALT) Concentrations
Time Frame: Week 48 and Week 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 37
international units per liter (IU/L)
  Week 48 | 62.6 (5.1)
  Week 72 | 64.5 (12.0)

7. Secondary Outcome: Percentage of HBeAg Negative Participants
Description: HBeAg seroconversion was defined as the absence of HBeAg (HBeAg negative) and the presence of anti-HBe (anti-HBe positive) for HBeAg positive participants. Percentage of HBeAg negative participants were reported.
Time Frame: Week 48 and Week 72
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 21
percentage of participants
  Week 48 (n= 20) | 25
  Week 72 (n= 21) | 29

8. Secondary Outcome: Percentage of Anti-HBe Positive Participants
Description: HBeAg seroconversion was defined as the absence of HBeAg (HBeAg negative) and the presence of anti-HBe (anti-HBe positive) for HBeAg participants. Percentage of Anti-HBe positive participants were reported.
Time Frame: Week 48 and Week 72
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 18
percentage of participants
  Week 48 (n= 17) | 41
  Week 72 (n= 18) | 33

ADVERSE EVENTS:
Time Frame: AEs were recorded from Screening till Week 72.
Description: All enrolled participants who received at least 1 dose of peginterferon alfa-2a were included in safety analysis.
Arm/Group | Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 15/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a (N=39)
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Subfebrile temperature (General disorders) | 1
Weakness (General disorders) | 1
Headache (General disorders) | 2
Anxiety (General disorders) | 1
Heartburn (General disorders) | 1
Arterial hypertension (Vascular disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Barrett esophagus (Gastrointestinal disorders) | 1
Stomach ache (Gastrointestinal disorders) | 1
Blood in stool (Gastrointestinal disorders) | 1
Prostate hyperplasia (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.